CLINICAL TRIAL: NCT01918969
Title: Determination of Reference Values of Circulating Endothelial Progenitor Cells CD34+144+CD14- and CD34+VEGF-R2+CD14- in a Blood Donnor Population
Brief Title: Reference Values of Circulating Endothelial Progenitor Cells
Acronym: ANOPEC2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hopital Jean Minjoz (Other)
Responsible Party: Principal Investigator, Prof. Sidney Chocron, MD, PhD, Hopital Jean Minjoz
Other Study IDs: 13/408
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Aortic Aneurysm
Keywords: Endothelial progenitor cells; Healthy blood donors
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood donors: Blood donors with no exclusion criteria i.e with a very low probability to have an aortic aneurysm

SUMMARY:
Circulating endothelial progenitor cells CD34+144+CD14- et CD34+VEGF-R2+CD14- have been shown to be inversely correlated to aortic aneurysm size. However reference values have not yet been determined. This study is aimed to determine reference values of CD34+144+CD14- et CD34+VEGF-R2+CD14- in healthy men and women blood donors.

DETAILED DESCRIPTION:
At the time of blood donation, 10mL of blood will be used to calculate the concentration of circulating endothelial progenitor cells CD34+144+CD14- et CD34+VEGF-R2+CD14- , and the ratio of circulating endothelial progenitor cells CD34+144+CD14- et CD34+VEGF-R2+CD14- / all circulating endothelial progenitor cells in order to determine reference values.

ELIGIBILITY:
Inclusion Criteria:

* Blood donors

Exclusion Criteria:

* age over 65
* Arterial hypertension (treated or not)
* Vascular disease
* smoker or former smoker who stopped smoking for less than a year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy blood donors
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Concentration of circulating endothelial progenitor cells CD34+144+CD14- and CD34+VEGF-R2+CD14- | 3 months

SECONDARY OUTCOMES:
Ratio of circulating endothelial progenitor cells CD34+144+CD14- et CD34+VEGF-R2+CD14- / all circulating endothelial progenitor cells | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Perrotti, MD, Principal Investigator — University of Franche-Comte; France; Pascal Morel, MD, PhD, Principal Investigator — Etablissement Français du Sang; Siamak Davani, MD, PhD, Study Chair — University of Franche-Comte. france
Locations (1):
- CHU Besançon, Besançon, France

REFERENCES:
- [Background] Parietti E, Pallandre JR, Deschaseaux F, Aupecle B, Durst C, Kantelip JP, Chocron S, Davani S. Presence of circulating endothelial progenitor cells and levels of stromal-derived factor-1alpha are associated with ascending aorta aneurysm size. Eur J Cardiothorac Surg. 2011 Jul;40(1):e6-12. doi: 10.1016/j.ejcts.2011.02.065. Epub 2011 Apr 9. PMID 21481600